CLINICAL TRIAL: NCT01706822
Title: Evaluating the Radial Reload Stapler With Tri-Staple TM Technology During Laparoscopic Low Anterior Resection for Rectal Cancer: A Prospective Multicenter Case Series
Brief Title: Radial Reload Laparoscopic LAR Case Series
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Medtronic - MITG (Industry)
Collaborators: University Hospitals Cleveland Medical Center (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVLARL0287
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Results first posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Covidien Radial Reload Stapler with Tri-Staple Technology (Experimental): Covidien Radial Reload Stapler with Tri-Staple Technology in laparoscopic LAR or proctosigmoidectomy
  Interventions: Device: Covidien Radial Reload Stapler with Tri-Staple Technology

INTERVENTIONS:
Device: Covidien Radial Reload Stapler with Tri-Staple Technology — Case series of patients arlaedy selected to undergo a laparoscopic LAR using the Radial Reload stapler

SUMMARY:
To evaluate the Radial Reload Stapler during laparoscopic low anterior resection (LAR) or anterior proctosigmoidectomy for rectal cancer by assessing the primary and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is able to understand and sign Informed Consent Form.
2. The subject is between 18-85 years of age.
3. The subject is anticipated to undergo a resection of the rectum with anastomosis below the peritoneal reflection.
4. The subject is anticipated to undergo mobilization and stapling of the rectum laparoscopically.

Exclusion Criteria:

1. Any female patient, who is pregnant, suspected pregnant, or nursing.
2. The participant is unable or unwilling to comply with the study requirements, follow-up schedule.
3. The participant has co-morbidities which, in the opinion of the investigator, will not be appropriate for the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Conor Delaney, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Covidien Radial Reload Stapler With Tri-Staple Technology: Covidien Radial Reload Stapler with Tri-Staple Technology in laparoscopic low anterior resection or proctosigmoidectomy.
Period: Overall Study
Arm/Group | Covidien Radial Reload Stapler With Tri-Staple Technology
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Covidien Radial Reload Stapler With Tri-Staple Technology
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: centimeters] | 165.0 (11.9)
Weight [Mean (Standard Deviation); unit: kilograms] | 73.9 (16.4)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 27.0 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: The Surgeon's Ability to Achieve a Staple Line at the Desired Level of the Rectum. The Reported Value Represents the Number of Participants in Whom the Criteria Was Met
Description: The surgeon's ability to achieve a staple line at the desired level of the rectum.
Time Frame: Operative
Measure: Number; unit: participants
Arm/Group | Covidien Radial Reload Stapler With Tri-Staple Technology
Number analyzed (Participants) | 8
participants | 6

2. Primary Outcome: The Ability to Achieve Adequate Distal Margins (Defined as >2cm [or >1cm With Clear Histologic Evaluation]) in the Low Rectum. The Reported Value Represents the Number of Participants in Whom the Criteria Was Met
Description: The ability to achieve adequate distal margins (defined as >2cm [or >1cm with clear histologic evaluation]) in the low rectum.
Time Frame: Operative
Measure: Number; unit: participants
Arm/Group | Covidien Radial Reload Stapler With Tri-Staple Technology
Number analyzed (Participants) | 8
participants | 7

3. Secondary Outcome: Access Measured by Surgeon Usability Questionnaire. The Reported Values Represent Percentage of Cases Surgeon Agree/Strongly Agree
Description: 1. Access measured by surgeon usability questionnaire.
Time Frame: Operatively
Measure: Number; unit: % of cases surgeon agree/strongly agree
Arm/Group | Covidien Radial Reload Stapler With Tri-Staple Technology
Number analyzed (Participants) | 8
% of cases surgeon agree/strongly agree
  Radial Reload (RR) easy to place in pelvis | 62.5
  RR was easy to get low in the pelvis | 87.5
  RR was easy to place in the colon and the rectum | 50
  Was the rectum contained in device after clamping | 50
  RR retained an adequate amount of tissue | 75
  Was the rectum transected with one firing | 12.5

4. Secondary Outcome: Visibility Measured by Surgeon Usability Questionnaire. The Reported Values Represent Percentage of Cases Surgeon Agree/Strongly Agree
Description: 2. Visibility measured by surgeon usability questionnaire
Time Frame: Operatively
Measure: Number; unit: % of cases surgeon agree/strongly agree
Arm/Group | Covidien Radial Reload Stapler With Tri-Staple Technology
Number analyzed (Participants) | 8
% of cases surgeon agree/strongly agree
  Visibility was adequate when RR was used | 87.5
  Did the instrument impede the visibility | 0

5. Secondary Outcome: Maneuverability Measured by Surgeon Usability Questionnaire. The Reported Values Represent Percentage of Cases Surgeon Agree/Strongly Agree
Description: 3. Maneuverability measured by surgeon usability questionnaire Question: Maneuverability of Radial reload during the procedure was adequate
Time Frame: Operatively
Measure: Number; unit: % of cases surgeon agree/strongly agree
Arm/Group | Covidien Radial Reload Stapler With Tri-Staple Technology
Number analyzed (Participants) | 8
% of cases surgeon agree/strongly agree | 62.5

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the 30 day follow-up visit
Arm/Group | Covidien Radial Reload Stapler With Tri-Staple Technology
Serious Adverse Events (participants affected / at risk) | 4/8
Other Adverse Events (participants affected / at risk) | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Covidien Radial Reload Stapler With Tri-Staple Technology (N=8)
Ileus (Gastrointestinal disorders) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Covidien Radial Reload Stapler With Tri-Staple Technology (N=8)
Urinary tract infection (Infections and infestations) | 1 (1)
Interoperative bleeding (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No